CLINICAL TRIAL: NCT05630079
Title: Short-term Variation of Atelectasis Score After High-frequency Percussions in Patients With Severe Acquired Brain Injury: a Retrospective Cohort Study.
Brief Title: Variation of Atelectasis Score After High-frequency Percussions in Severe Acquired Brain Injury
Status: Completed | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Paolo Banfi, Head of Pneumological Rehabilitation, Fondazione Don Carlo Gnocchi Onlus
Other Study IDs: FDG_05_17/02/2021
Record Dates: First submitted 2022-09-26; First posted 2022-11-29 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Atelectasis; Acquired Brain Injury; Respiratory Rehabilitation
MeSH Terms: conditions — Pulmonary Atelectasis; Brain Injuries | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Metaneb®: Patients admitted for severe acquired brain injury (sABI) in Neurological Rehabilitation Unit of IRCCS "Santa Maria Nascente - Fondazione Don Gnocchi" received the MetaNeb® system treatment. It consist of simultaneous combination of positive pressure, continuous high frequency oscillations and aerosol delivery
  Interventions: Device: Treatment with Metaneb®
- IPV®: Patients with severe acquired brain injury from Neurological Rehabilitation Unit of IRCCS Fondazione Don Gnocchi, S.M. Nascente received the IPV® treatment. The principle of IPV® is to open collapsed airways and mobilize intrabronchial secretions through the delivery of small tidal volume at high frequency. IPV® adjusts the percussions to the changes in the mechanical properties of the patient's respiratory system: in case of high resistance, it produces small tidal volume at high pressure and low frequency; vice versa in case of low resistance, it produces large tidal volume at low pressure and high frequency
  Interventions: Device: Treatment with IPV®

INTERVENTIONS:
Device: Treatment with Metaneb® — Every patient of this group receive 3 daily treatments of 20 minutes each, performed at approximately 4-hour intervals.
  Each treatment with MetaNeb system consists of four cycles: : 5 minutes of Continuous Positive Expiratory Pressure (CPEP) for lung re-expansion (Cycle I), 5 minutes of Chest High Frequency Oscillation (CHFO) for secretion clearance (Cycle II), 5 min of CPEP (Cycle III), 5 minutes of CHFO (Cycle IV). Treatments are performed by respiratory physiotherapists and the pressure setted was the highest tolerated by the patient. It's associated with the administration of aerosols with 10 ml of saline solution 0.9% and are carried out by connecting the tracheostomy cannula cuffed to the catheter mount.
  Groups: Metaneb®
Device: Treatment with IPV® — Each treatment with IPV provides 3 daily treatments of 20 minutes with the high percussion frequency tolerated by the patient. and I/E ratio: 1/1.2. Treatments are performed by respiratory physiotherapists and the pressure setted was the highest tolerated by the patient. It is associated with the administration of aerosols with 10 ml of saline solution 0.9% [-] and are carried out by connecting the tracheostomy cannula cuffed to the catheter mount.
  Groups: IPV®

SUMMARY:
Investigators conduced in the Neurological Rehabilitation Unit of the IRCCS "S.Maria Nascente - Fondazione Don Gnocchi", (Milan) a retrospective study on 19 patients hospitalized between September 2018 and February 2021, with the aim of comparing the efficacy of the two devices, MetaNeb® and Intrapulmonary Percussion Ventilation (IPV®).

The efficacy was evaluated considering the change of various measures after two weeks of treatment. The main outcome considered is the atelectasis score, assigned by two radiologists who blindly and retrospectively evaluated it on high-resolution computed tomography (HRTC) images

DETAILED DESCRIPTION:
Patients with severe acquired brain injury (sABI) frequently exhibit pulmonary complications, with atelectasis and/or consolidation of the lower lobes. The atelectasis in critically ill patients is a risk factor for pneumonia and increase the possibility to develop dysventilation syndrome with consequent negative impacts on gas exchanges.

To the best of our knowledge, there is no study investigating the use of the two devices for the treatment of atelectasis in the specific population of non-cooperative tracheostomized patients with sABI who had been spontaneously breathing with no mechanical ventilation support.

ELIGIBILITY:
Inclusion Criteria:

* Spontaneous breathing 24h/24h
* Presence of tracheostomy cannula
* Presence of atelectasis diagnosed through High Resolution Computed Tomography
* Levels of Cognitive Functioning (LCF) ≤ 5
* No pneumothorax
* Consent signed

Exclusion Criteria:

* Age under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted for severe acquired brain injury (sABI) in Neurological Rehabilitation Unit of IRCCS "Santa Maria Nascente - Fondazione Don Gnocchi" from September 2018 to February 2021
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2022-02-22 (Actual)

PRIMARY OUTCOMES:
Variation of atelectasis score after treatment | 15 days
  The aim is to compare the effect of the two devices, IPV® and MetaNeb® in the treatment of atelectasis. The atelectasis score is assigned by two radiologists who blindly and retrospectively evaluated it on high-resolution computed tomography (HRTC) images
Automatic score by Siemens | 15 days
  Comparing the atelectasis score using an automatic score generated by Siemens (syngo.via CT Pneumonia Analysis), in case of discrepancy between all radiologists

SECONDARY OUTCOMES:
Blood Gas Analysis | 15 days
  Changes of respiratory parameters in terms of normalization of oxyemia (Arterial Pressure of oxygen 80-100 mmHg) and normalization of capnia (Arterial Pressure of carbon dioxide 35-45 mmHg), assessed by blood gas analysis
Peripheral Oxygen Saturation (SpO2) at night | 15 days
  Average SpO2, Lowest SpO2, <90% (lenght of time SpO2 dropped below 90%), Average Heart Rate

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Santa Maria Nascente, Fondazione Don Gnocchi, Milan, Italy